CLINICAL TRIAL: NCT04342572
Title: Intra-arterial Chemotherapy for Retinoblastoma (IAC)
Brief Title: Intra-arterial Chemotherapy for Retinoblastoma
Acronym: IAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202006160
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-arterial injections of melphalan (Experimental): -Participants will receive intra-arterial injections of melphalan Q4W for 3 cycles.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — -The drug is commerically available
  Other Names: Evomela

SUMMARY:
Children with retinoblastoma who may benefit from intra-arterial chemotherapy will receive up to 3 doses of melphalan and will be assessed for feasibility, toxicity, and response.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with retinoblastoma >4 months of age16
* Patients whose other treatment options would require systemic chemotherapy, radiotherapy, or enucleation
* Patient or parent/legal guardian must sign a written informed consent
* One of a, b, or c:

  * Patients who have bilateral COG stage B, C, D, or E retinoblastoma (refer to Appendix A) who have undergone systemic chemotherapy without resolution (meaning either has not had CR or has progressed despite systemic chemotherapy) and would have the following treatment options remaining:

    * IAC
    * enucleation of one eye
    * local radiation
  * Patients with non-germline retinoblastoma with unilateral disease who have COG A, B, C, or D tumors (refer to Appendix A).
  * Other patients may be considered on a case by case basis after discussion with pediatric ophthalmology, hematology/oncology, and interventional neuroradiology.

Exclusion Criteria:

* Opaque or hazy media which precluded visualization of the fundus.
* New or recurrent retinoblastoma that can be controlled with other conservative measures such as cryotherapy, thermotherapy, or plaque radiotherapy.
* Unilateral COG group E retinoblastoma (refer to Appendix A) with very poor visual prognosis as defined by pediatric ophthalmologist.
* Patients who would benefit from systemic chemotherapy.
* Patients with clinical or radiological evidence suggestive of retinoblastoma invasion of the optic nerve, choroid, sclera, orbit or metastatic sites.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Participants of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of intra-arterial chemotherapy as measured by the number of participants who receive 3 intra-arterial injections of melphalan | Completion of enrollment and treatment of all patients (estimated to be 32 months)
  -Feasibility is defined as the ability to receive 3 intra-arterial injections of melphalan per patient.

SECONDARY OUTCOMES:
Rate of procedure-related complications | Through 30 days following completion of treatment (estimated to be 4 months)
Rate of ocular salvage | 2 years post-treatment
  A patient will be considered a successful ocular salvage if the child does not experience enucleation because of disease progression or toxicity during 2 years of follow-up.
Visual acuity as measured by Cardiff testing | 6 months post-treatment
Rate of metastatic disease | Completion of treatment (estimated to be 3 months)
  -Patients will be determined to have metastatic disease if they have received 1 or more administrations of IAC and they are found to have progression of disease or appearance of tumor outside of the eye after protocol therapy. Pineal tumors will not be considered metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Reynolds, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine (Saint Louis Children's Hospital), St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu